CLINICAL TRIAL: NCT04663672
Title: Placebo-Controlled, Randomized, Double-Blind Study of the Efficacy of Targeted Memory Reactivation for Enhancing Exposure Therapy
Brief Title: Efficacy of Targeted Memory Reactivation for Enhancing Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Prinicipal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-09-0058
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Claustrophobia; Obsessive-Compulsive Disorder; Arachnophobia
Keywords: Targeted Memory Reactivation; Memory Consolidation; Exposure Therapy; Sleep
MeSH Terms: conditions — Claustrophobia; Obsessive-Compulsive Disorder; Arachnophobia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure Therapy + Exposure Scent Cue During Sleep (Experimental): Participants will undergo exposure treatment for their target fear while in the presence of a distinctive odor. Exposure will occur in repeated 4-minute trials. Exposure will continue for 40 minutes or until peak fear decreases by at least 35 points on a 100 point scale, compared to peak fear during the initial trial. Participants will subsequently sleep in the presence of the exposure scent.
  Interventions: Other: Experimental Scent; Behavioral: In-Vivo Exposure
- Exposure Therapy + Novel Scent During Sleep (Placebo Comparator): Participants will undergo exposure treatment for their target fear while in the presence of a distinctive odor. Exposure will occur in repeated 4-minute trials. Exposure will continue for 40 minutes or until peak fear decreases by at least 35 points on a 100 point scale, compared to peak fear during the initial trial. Participants will subsequently sleep in the presence of a novel scent.
  Interventions: Other: Control Scent; Behavioral: In-Vivo Exposure
- Exposure Therapy + No-Scent Control During Sleep (Sham Comparator): Participants will undergo exposure treatment for their target fear while in the presence of a distinctive odor. Exposure will occur in repeated 4-minute trials. Exposure will continue for 40 minutes or until peak fear decreases by at least 35 points on a 100 point scale, compared to peak fear during the initial trial. Participants will subsequently sleep in the presence of an odorless control vehicle.
  Interventions: Other: No-Scent Control; Behavioral: In-Vivo Exposure

INTERVENTIONS:
Other: Experimental Scent — Participants will sleep in the presence of the exposure scent, delivered by an Airwick Essential Oils diffuser
  Arms: Exposure Therapy + Exposure Scent Cue During Sleep
Other: Control Scent — Participants will sleep in the presence of a novel scent, delivered by an Airwick Essential Oils diffuser
  Arms: Exposure Therapy + Novel Scent During Sleep
Other: No-Scent Control — Participants will sleep in the presence of an odorless control vehicle, delivered by an Airwick Essential Oils diffuser
  Arms: Exposure Therapy + No-Scent Control During Sleep
Behavioral: In-Vivo Exposure — Participants will receive 40 minutes of in-vivo exposure therapy to feared targets in the presence of a distinctive exposure scent.

SUMMARY:
This study evaluates whether a scent applied during exposure therapy and during subsequent sleep will increase the durability of treatment effects for individuals with fear of spiders, contamination, and enclosed spaces.

DETAILED DESCRIPTION:
Newly acquired memories encoded during wakefulness are spontaneously re-activated during sleep, resulting in synaptic potentiation and strengthening of the re-activated traces. Targeted memory reactivation (TMR) typically involves a period of initial learning in the presence of an olfactory or auditory contextual cue, coupled with later presentation of the cue during sleep to ostensibly facilitate memory reactivation and consolidation. Numerous studies have found evidence of improved task performance subsequent to cue-induced neuronal replay, however application of TMR to treatment of naturally acquired, clinically significant fear has been limited.

The present study will will provide a rigorous test of TMR's efficacy as an augmentative strategy for exposure therapy. It is hypothesized that participants who sleep in the presence of the same odor that they are exposed to during exposure therapy will exhibit reduced fear at follow up, relative to participants who sleep in the presence of a different odor, or a non-odorous control.

ELIGIBILITY:
Inclusion Criteria:

* Marked anxiety in at least one fear domain (spiders, contamination, or enclosed spaces), as determined by the presence of both:

  1. self-reported peak anxiety of at least 50 on a 100 point scale in response to two behavioral approach tasks
  2. self-report measures meeting the following cutoffs for the target fear:
* Fear of Spiders Questionnaire ≥ 50
* Obsessive-Compulsive Inventory-Revised (Washing Subscale) ≥ 4
* Claustrophobia Screener ≥ 2

Exclusion Criteria:

* Diagnosed sleep disorder
* Current sleep medication usage
* Inability to differentiate two different odors from an indoor scent diffuser
* Current psychotherapy for fear of spiders, snakes, enclosed spaces, or contamination
* Current use of air fresheners, scented candles, or other items with odors related to those used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in fear response during two behavioral approach tasks across time points | Baseline (Day 1); Post-treatment (Day 1; immediately after treatment); One Week Follow-Up (Day 8; one week after treatment); One Month Follow-Up (Day 31; one month after treatment)
  Change in subjective units of distress (0 = no fear, to 100 = extreme fear) and skin conductance in response to approaching a feared stimulus, from baseline to one month follow-up

SECONDARY OUTCOMES:
Change in arachnophobia symptom severity across time-points | Baseline (Day 1); One Week Follow-Up (Day 8; one week after treatment); One Month Follow-Up (Day 31; one month after treatment)
  Change in total score on the Fear of Spiders Questionnaire from baseline to one month follow-up
Change in claustrophobia symptom severity across time points | Baseline (Day 1); One Week Follow-Up (Day 8; one week after treatment); One Month Follow-Up (Day 31; one month after treatment)
  Change in total score on the Claustrophobia Questionnaire from baseline to one month follow-up
Change in contamination fear symptom severity across time points | Baseline (Day 1); One Week Follow-Up (Day 8; one week after treatment); One Month Follow-Up (Day 31; one month after treatment)
  Change in total score on the contamination subscale of the Padua Inventory- Washington State University Revision from baseline to one month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for the Study of Anxiety Disorders, University of Texas at Austin, Austin, Texas, United States